CLINICAL TRIAL: NCT02945150
Title: A Proof of Concept Study of Preemptive Treatment With Grazoprevir and Elbasvir for Donor HCV Positive to Recipient HCV Negative Kidney Transplant
Brief Title: Preemptive Treatment With Grazoprevir and Elbasvir for Donor HCV Positive to Recipient HCV Negative Kidney Transplant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Raymond Chung, Director, Hepatology, Massachusetts General Hospital, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016P002051; Merck MISP 54841 (Other Grant/Funding Number: Merck)
Record Dates: First submitted 2016-10-21; First posted 2016-10-26 (Estimated); Results first posted 2020-02-26 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Renal Failure
Keywords: hemodialysis; peritoneal dialysis; renal failure; kidney transplant
MeSH Terms: conditions — Renal Insufficiency | interventions — elbasvir; grazoprevir; elbasvir-grazoprevir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Elbasvir/grazoprevir for HCV+ kidney transplant recipients (Experimental): Elbasvir (50mg) / grazoprevir (100mg) (fixed dose combination) treatment for Hepatitis C virus (HCV)-naive recipients who receive a kidney transplant from a deceased, HCV-infected donor
  Subjects receive first dose on-call to operating room, and continue daily for 12 weeks. Treatment length is extended to 16 weeks and ribavirin (daily dose 1000 mg for those <75 kg and 1200 mg for those ≥75 kg) if subject receives a kidney from a donor who is infected with HCV containing resistance-associated variants (RAV).
  Interventions: Drug: elbasvir (50mg) / grazoprevir (100mg) (fixed dose combination)

INTERVENTIONS:
Drug: elbasvir (50mg) / grazoprevir (100mg) (fixed dose combination) — Elbasvir (50mg) / grazoprevir (100mg) (fixed dose combination) treatment for Hepatitis C virus (HCV)-naive recipients who receive a kidney transplant from a deceased, HCV-infected donor
  Subjects receive first dose on-call to operating room, and continue daily for 12 weeks. Treatment length is extended to 16 weeks and ribavirin (daily dose 1000 mg for those <75 kg and 1200 mg for those ≥75 kg) if subject receives a kidney from a donor who is infected with HCV containing resistance-associated variants (RAV).
  Other Names: Zepatier

SUMMARY:
Proof of concept, open-label single center study for the donation of HCV positive kidneys to HCV negative patients, with preemptive, interventional treatment to prevent HCV transmission upon transplantation.

DETAILED DESCRIPTION:
The study objective is to determine if the administration of grazoprevir and elbasvir (with or without ribavirin) for 12-16 weeks after kidney transplantation prevents the spread of HCV infection from a donor kidney with known HCV genotype 1 or 4 infection to a HCV negative recipient as evidenced by a negative HCV viral RNA at 12 weeks post treatment

ELIGIBILITY:
Inclusion Criteria:

1. Must meet Massachusetts General Hospital (MGH) transplant center criteria and already be listed for isolated kidney transplant
2. No available living kidney donor
3. Has ≤ 730 days (two years) of accrued transplant waiting time if blood type A and ≤ 1095 days of accrued transplant waiting time if blood type B or O.
4. On chronic hemodialysis or peritoneal dialysis or has a glomerular filtration rate <15mL/min/1.73m2 at the time of screening
5. Weight ≥ 50kg
6. Serum alanine transaminase (ALT) within normal limits

Exclusion Criteria:

1. AB blood type
2. Body mass index (BMI > 35
3. History of liver disease
4. Pregnant or nursing (lactating) women
5. Cardiomyopathy (LV ejection fraction < 50%)
6. Positive crossmatch or positive donor specific antibodies
7. Human immunodeficiency virus (HIV) positive
8. Hepatitis C virus (HCV) RNA positive
9. Hepatitis B virus (HBV) surface antigen positive
10. Any contraindication to kidney transplant per MGH center protocol

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2020-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Chung, MD, Principal Investigator — Massachusetts General Hospital (Partners Healthcare)
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with study sponsor and with the hopes of publication.
Supporting Information: Study Protocol
Time Frame: Protocol will be shared for up to 1 year after the final patient has dosed.
Access Criteria: Protocol will only be shared with Institutional Review Board (IRB) approved study staff and PI approved collaborators.

REFERENCES:
- [Background] Kucirka LM, Singer AL, Ros RL, Montgomery RA, Dagher NN, Segev DL. Underutilization of hepatitis C-positive kidneys for hepatitis C-positive recipients. Am J Transplant. 2010 May;10(5):1238-46. doi: 10.1111/j.1600-6143.2010.03091.x. Epub 2010 Mar 26. PMID 20353475

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 33 patients signed consent for the study. Of those, 23 patients were deemed "ready" for transplant and were put on the waitlist for a HCV kidney (10 patients did not meet the "readiness" criteria for kidney transplantation). Of those, 8 patients were transplanted with an HCV+ kidney.
Period: Overall Study
Arm/Group | Elbasvir/Grazoprevir for HCV+ Kidney Transplant Recipients
Started | 8
SVR12 | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Elbasvir/Grazoprevir for HCV+ Kidney Transplant Recipients
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
End stage renal disease (ESRD) cause [Count of Participants; unit: Participants]
  Diabetes/hypertension | 3
  IgA nephropathy | 3
  Polycystic kidney disease | 1
  Systemic lupus erythematosus | 1
Blood type [Count of Participants; unit: Participants]
  A | 5
  O | 3
Prior transplant [Count of Participants; unit: Participants] | 1
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 29.9 [28 to 31.6]
History of diabetes [Count of Participants; unit: Participants] | 4
Days on waitlist prior to consent [Median (Inter-Quartile Range); unit: days] | 482.5 [367.25 to 625.25]
Days from consent to transplant [Median (Inter-Quartile Range); unit: days] | 207.5 [86.75 to 426.75]
Length of hospital stay [Count of Participants; unit: Participants]
  4 days | 2
  5 days | 3
  6 days | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Undetectable HCV RNA at SVR12
Description: Sustained virologic response at 12-weeks post-treatment (SVR12), as defined by negative HCV viral load, after 12-16 weeks of elbasvir/grazoprevir treatment in patients who receive a kidney transplant from a deceased donor infected with HCV.
Time Frame: 12 weeks post-treatment (24 weeks post-transplant)
Measure: Count of Participants; unit: Participants
Arm/Group | Elbasvir/Grazoprevir for HCV+ Kidney Transplant Recipients
Number analyzed (Participants) | 8
Participants | 8

2. Secondary Outcome: Number of Subjects With Undetectable Serum HCV RNA at Study Day 7, 14, 28, 56, 84, 112, 168, 252, 365
Description: Subjects had Hepatitis C viral load assessed at each study visit. Here we looked at the proportion of subjects with undetectable serum HCV RNA at study day 7, 14, 28, 56, 84, 112, 168, 252, 365.
Time Frame: 1 year post transplant
Population: Patients who received a HCV+ kidney transplant and were treated with elbasvir (50mg) / grazoprevir (100mg) for 12 weeks following transplant.
Measure: Number; unit: participants
Arm/Group | Elbasvir/Grazoprevir for HCV+ Kidney Transplant Recipients
Number analyzed (Participants) | 8
participants
  Day 7 | 7
  Day 14 | 8
  Day 28 | 8
  Day 56 | 8
  Day 84 | 8
  Day 112 | 8
  Day 168 | 8
  Day 252 | 8
  Day 365 | 8

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from time of consent to 1 year post-transplant
Description: Adverse event data collection is still ongoing for two participants who have yet to reach the one year-post transplant mark.
Arm/Group | Elbasvir/Grazoprevir for HCV+ Kidney Transplant Recipients
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 4/8
Other Adverse Events (participants affected / at risk) | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elbasvir/Grazoprevir for HCV+ Kidney Transplant Recipients (N=8)
Lymphocele (Surgical and medical procedures) | 1 (1) — Lymphocele post kidney transplant requiring drain placement, and subsequent laparoscopic fenestration of peri-nephric lymphocele (x2).
Renal vein thrombosis (Renal and urinary disorders) | 1 (1) — Immediate graft failure due to renal vein thrombosis. Allograft explanted on post-operative day 1. Patient anticoagulated and returned to dialysis. Workup for coagulopathy demonstrated positive test for lupus anticoagulant. Achieved SVR12.
Delayed graft function (Renal and urinary disorders) | 1 (1) — Patient readmitted to hospital for one day for delayed graft function. Graft function improved and patient was discharged.
Acute kidney injury (AKI) (Renal and urinary disorders) | 1 (1) — Admitted to hospital for AKI. Discharged after one day upon improvement.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elbasvir/Grazoprevir for HCV+ Kidney Transplant Recipients (N=8)
Elevated alanine transaminase (ALT) (Hepatobiliary disorders) | 3 (8) — ALT measured at baseline, day 1, day 3, day 7, day 14, day 28, day 42, day 56, day 70, day 84, day 112, day 168, day 252, and day 365 High ALT defined as being above 55 U/L for males and 33 U/L for females
Elevated aspartate transaminase (AST) (Hepatobiliary disorders) | 3 (8) — AST measured at baseline, day 1, day 3, day 7, day 14, day 28, day 42, day 56, day 70, day 84, day 112, day 168, day 252, and day 365 High AST defined as being above 40 U/L for males and 32 U/L for females
Elevated total bilirubin (Hepatobiliary disorders) | 1 (1) — Bilirubin measured at baseline, day 1, day 3, day 7, day 14, day 28, day 42, day 56, day 70, day 84, day 112, day 168, day 252, and day 365 High bilirubin defined as being above 1.0 mg/dL
Diarrhea (Gastrointestinal disorders) | 1 (1) — Patient who was admitted for AKI also had diarrhea during admission. Was discharged after 1 day upon improvement.
Abdominal pain (Gastrointestinal disorders) | 1 (1) — Patient who was admitted for AKI also had abdominal pain during admission. Was discharged after 1 day upon improvement.
Hematoma at surgical site (Surgical and medical procedures) | 1 (1) — Patient who was admitted for AKI also had hematoma at surgical site during admission. Was discharged after 1 day upon improvement.
Hypophosphatemia (Blood and lymphatic system disorders) | 1 (1) — Patient who was admitted for AKI also had hypophosphatemia during admission. Was discharged after 1 day upon improvement.
Hypomagnesemia (Blood and lymphatic system disorders) | 1 (1) — Patient who was admitted for AKI also had hypomagnesemia during admission. Was discharged after 1 day upon improvement.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT02945150/Prot_SAP_000.pdf